CLINICAL TRIAL: NCT01841372
Title: A Virtual Reality Intervention (Second Life) to Improve Weight Maintenance
Brief Title: A Virtual Reality Intervention to Improve Weight Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Donnelly, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13610
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Weight Loss
Keywords: Obesity; Overweight; Weight Maintenance
MeSH Terms: conditions — Weight Loss; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Phone Conference Call (Active Comparator): Group phone clinic will be conducted weekly during the first 9 months and twice/month during the final 9 months (3 to 12 months).
  Interventions: Behavioral: Group Phone Conference Call
- Second Life (2L) (Experimental): 2L group meeting will be conducted weekly during the first 9 months and twice/month during the final 9 months
  Interventions: Other: Second Life

INTERVENTIONS:
Other: Second Life — Second Life is an online virtual reality environment.
  Arms: Second Life (2L)
Behavioral: Group Phone Conference Call
  Arms: Group Phone Conference Call

SUMMARY:
The purpose of this study is to determine if use of a virtual reality platform, Second Life, is more effective than traditional face-to-face methods for maintaining weight loss in overweight and obese individuals.

DETAILED DESCRIPTION:
This study has two main parts. During the first 6 months (-6 to 0 months)potential subjects will be on a diet developed by researchers at the University of Kansas Medical Center (KUMC). Subsequent to 6 months, participants who lost 5% weight will begin the weight maintenance phase of the study (0-12 months). Thus the total duration of the study is 18 months.

Approximately 68% of U.S. adults are classified as overweight or obese (BMI >25). Behaviorally based weight loss programs, typically delivered by face-to-face clinics, produce clinically significant reductions in body weight over 3-6 months. However, approximately 50% of those who lose weight regain more than 45-75% of the weight lost within 12-30 months. Face-to-face clinics present many barriers and burdens to individuals including scheduling and logistical and financial burdens.

Virtual Reality (VR) environments allow participants to create virtual representations of themselves called "avatars". An existing VR called "Second Life" will be used for participants randomized to VR. Participants avatars attend group meetings and use headsets for voice communication to interact with each other.

Those not randomized to VR will participate in traditional face-to-face group weight loss intervention. The study will examine many different factors to determine if those participants in the Second Life group experience improved weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with a BMI of 25 to 39.9 kg/m2
* Able to obtain clearance for participation from their primary care physician (PCP)
* Have access to a computer with internet that meets Second Life system requirements

Exclusion Criteria:

* Report participating in a research project involving weight loss or PA in the previous 6 months
* Report a regular exercise or PA program
* Not weight stable (+/-2.27 kg) for 3 months prior to intake
* Unwilling to be randomized to phone or 2L clinics subsequent to weight loss
* Report being pregnant during the previous 6 months, lactating, or planned pregnancy in the following 18 months
* Report serious medical risk such as type 1 diabetes, cancer, recent cardiac event (i.e. heart attack, angioplasty, etc.)
* Report eating disorders as determined by the Eating Attitudes Test using a score of 20 or greater
* Report current treatment for psychological issues, or taking psychotropic medications
* Report adherence to specialized diet regimes, i.e., multiple food allergies, vegetarian, macrobiotic, etc.
* Do not have access to grocery shopping and meal preparation (i.e. Military, college cafeteria plan, etc.).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Difference in Weight Change | Change from month 0 (after 6 mo weight loss) to Month 12
  Weight change measured during Month 0 (after 6 mo weight loss) to Month 12.

SECONDARY OUTCOMES:
Total Attendance at Meetings | Month 0 to12 Months
  Number of times each individual attended group meeting during the course of the weight maintenance phase.
Assessment of Self-Efficacy for Weight Loss | Change from Month 0 to 12 Months
  Weight loss self-efficacy will be assessed using the Weight Efficacy Lifestyle Questionnaire. This scale assess overeating in tempting situations. Participants rate their level of confidence on a 10-point Likert-scale with higher values indicating greater confidence to resist overeating.
Assessment of Self-Efficacy for Physical Activity (PA) | Change from Month 0 to 12 Months
  Physical activity self-efficacy will be assessed using the 5-item exercise self-efficacy scale. Participants rate their confidence level (1 = not confident at all to 7 = very confident) to engage in PA in a number of different situations including making time for exercise, resisting lapse, etc.
Assessment of Self-Efficacy for Problem Solving Skills | Change from Month 0 to 12 Months
  Problem-solving abilities will be assessed using the Social Problem Solving Inventory-Revised, short form (SPSI-R:S). The SPSI-R:S is a 25-item instrument with five component scales to assess problem-solving styles and solution generation.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, Ed.D., Principal Investigator — University of Kansas Medical Center; Debra Sullivan, PhD, RD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Sullivan DK, Goetz JR, Gibson CA, Mayo MS, Washburn RA, Lee Y, Ptomey LT, Donnelly JE. A virtual reality intervention (Second Life) to improve weight maintenance: Rationale and design for an 18-month randomized trial. Contemp Clin Trials. 2016 Jan;46:77-84. doi: 10.1016/j.cct.2015.11.019. Epub 2015 Nov 23. PMID 26616535